CLINICAL TRIAL: NCT04743466
Title: Evaluation of a Causal Association Between Testosterone Levels, Dementia, and Adverse Mental Health Outcomes: A Mendelian Randomization Analysis
Brief Title: Evaluation of Association Between Testosterone Levels, Dementia, and Adverse Mental Health Outcomes
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1061; NCI-2020-13782 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1061 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Disorder; Depression; Genetic Disorder; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Anxiety Disorders; Depression; Genetic Diseases, Inborn; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biobank review): Patients' records from institutional or national biobanks are reviewed.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Biobank records are reviewed

SUMMARY:
This study evaluates the association between testosterone levels and risk of dementia and adverse mental health outcomes (e.g. depression and anxiety). It is not known whether low testosterone levels may be associated with an increased risk of dementia. Learning about the association between testosterone levels and risk of dementia may help determine the long-term effects of androgen deprivation therapy and may help improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To use a Mendelian randomization study design to determine whether genetically predicted decreased testosterone levels are associated with an increased risk of dementia.

SECONDARY OBJECTIVE:

I. To examine whether genetically predicted decreased testosterone levels are associated with worse cognitive function and adverse mental health outcomes.

OUTLINE:

Patients' records from institutional or national biobanks are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Have volunteered to participate in institutional or national biobanks, mainly the UK Biobank and the Kaiser Permanente Research Bank, and those that have previously participated in studies that resulted in de-identified clinical and genetic data being make available on public archives, mainly the database of Genotypes and Phenotypes (dbGaP)
* No special populations (adults unable to consent, individuals not yet adults, pregnant women, or prisoners)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals have volunteered to participate in institutional or national biobanks
Sampling Method: Non-Probability Sample
Enrollment: 700000 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Association between germline genetic predictors (single nucleotide variants) of lower testosterone levels and dementia risk | Up to 2 years
  Will utilize genetic variants associated with testosterone levels at genome-wide statistical significance thresholds (P < 5 x 10-8) in published meta-analyses. Will additionally conduct a genome-wide association study with testosterone values in the UK Biobank. Will construct a weighted genetic risk score based on the strength of each variant's association with testosterone levels in published datasets. The results of the weighted method will be scaled per standard deviation (SD) of testosterone levels so that effect sizes represent the odds ratio of the outcome (e.g. dementia) per genetically predicted SD decrease in testosterone levels. Will also utilize risk scores with less stringent significance thresholds in secondary analyses (P < 5 x 10-6).

SECONDARY OUTCOMES:
Depression | Up to 2 years
  Association between low testosterone levels and depression will be examined. Will construct a weighted genetic risk score based on the strength of each variant's association with testosterone levels in published datasets. The results of the weighted method will be scaled per standard deviation (SD) of testosterone levels so that effect sizes represent the odds ratio of the outcome (e.g. dementia) per genetically predicted SD decrease in testosterone levels. Will also utilize risk scores with less stringent significance thresholds in secondary analyses (P < 5 x 10-6).
Anxiety | Up to 2 years
  Association between low testosterone levels and anxiety will be examined. Will construct a weighted genetic risk score based on the strength of each variant's association with testosterone levels in published datasets. The results of the weighted method will be scaled per standard deviation (SD) of testosterone levels so that effect sizes represent the odds ratio of the outcome (e.g. dementia) per genetically predicted SD decrease in testosterone levels. Will also utilize risk scores with less stringent significance thresholds in secondary analyses (P < 5 x 10-6).
Cognitive/mental health | Up to 2 years
  Association between low testosterone levels and cognitive/mental health will be examined. Will construct a weighted genetic risk score based on the strength of each variant's association with testosterone levels in published datasets. The results of the weighted method will be scaled per standard deviation (SD) of testosterone levels so that effect sizes represent the odds ratio of the outcome (e.g. dementia) per genetically predicted SD decrease in testosterone levels. Will also utilize risk scores with less stringent significance thresholds in secondary analyses (P < 5 x 10-6).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Nead, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States